CLINICAL TRIAL: NCT01941576
Title: Effects of rhBNP in Pediatrics After Corrective Repair of Tetralogy Of Fallot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xu Zhuoming, Vice Chief, Department of thoracic and cardiovascular surgery, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SJTUMS-20130903
Record Dates: First submitted 2013-09-03; First posted 2013-09-13 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Congenital Heart Defects; Tetralogy Of Fallot
Keywords: Heart defects, Congenital; rhBNP; heart failure
MeSH Terms: conditions — Heart Defects, Congenital; Tetralogy of Fallot; Heart Failure | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rhBNP Group (Experimental): Patients after corrective repair of Tetralogy Of Fallot will be treat with routinely therapy, including inotropics and diuretics, combined a rhBNP infusion 24 hours after operation. The dose of recombinant human brain natriuretic peptide (rhBNP) will be 1.5 mcg/kg for loading, followed by continuous infusion recombinant human brain natriuretic peptide 0.01-0.01mcg/kg/min for 72 hours.
  Interventions: Drug: recombinant human brain natriuretic peptide (rhBNP)
- Placebo Group (Placebo Comparator): Patients after corrective repair of Tetralogy Of Fallot will be treat with routinely therapy, including inotropics and diuretics, combined a placebo infusion 24 hours after operation.
  Interventions: Drug: Placebo (0.9% sodium chloride)

INTERVENTIONS:
Drug: recombinant human brain natriuretic peptide (rhBNP) — Patients are first given a loading dose of recombinant human brain natriuretic peptide (rhBNP) 1.5 mcg/kg, followed by continuous infusion recombinant human brain natriuretic peptide 0.01-0.01mcg/kg/min for 72 hours.
  Arms: rhBNP Group
Drug: Placebo (0.9% sodium chloride) — Patients after corrective repair of Tetralogy Of Fallot will be treat with routinely therapy, including inotropics and diuretics, combined a placebo infusion 24 hours after operation.
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to determine the effects of rhRNP on urine output and hemodynamics following corrective repair of Tetralogy Of Fallot.

DETAILED DESCRIPTION:
CVP(central venous pressure) and cardiac output are serious index in children with Tetralogy Of Fallot after the corrective repair.The purpose of this study is to investigate if the therapy of rhRNP can improve the survival and life quality after the corrective repair of Tetralogy Of Fallot.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained from patient's legally acceptable representative.
* Pediatric patients after Repair of Tetralogy Of Fallot.

Exclusion Criteria:

* Psychotic, addictive or other disorder limiting the ability to provide informed consent or to comply with study requirements.
* Treatment or planned treatment with another investigational drug within 3 months of screening.
* Known hypersensitivity to bosentan or any of the excipients
* cardiogenic shock and inclination of hypotension（SBP< 60mmHg）.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline in BNP and CVP after the infusion of rhBNP | 12 months after operation of Tetralogy Of Fallot
  we will evaluate the cardiac function through the consecutive changed numerical value of brain natriuretic peptide and Central Venous Pressure.

SECONDARY OUTCOMES:
Changes from baseline on the volume of urine out and numerical value of serum creatinine and blood urea nitrogen | 12 months after operation of Tetralogy Of Fallot
  we evaluate the renal function through the volume of urine out and numerical value of serum creatinine and blood urea nitrogen.

CONTACTS AND LOCATIONS:
Overall Officials: Zhuoming Xu, MD,PhD, Study Director — Shanghai Children's Medical Center
Locations (1):
- Cardiac intensive care unit, Department of cardiothoracic vascular surgery, Shanghai Children's Medical Center, Medical college of Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China